CLINICAL TRIAL: NCT06507852
Title: Retrospective Assessment of Inclisiran Adherence, Treatment Patterns, Patient Characteristics, and Effectiveness Among ASCVD Patients With Hypercholesterolemia, ASCVD-risk Equivalent Patients With Hypercholesterolemia and Familial Hypercholesterolemia Patients Prescribed LEQVIO® (Inclisiran) in a Real-world Setting
Brief Title: A Real-world Study of Inclisiran Adherence, Treatment Patterns, Patient Characteristics, and Effectiveness in ASCVD Patients With Hypercholesterolemia, ASCVD-risk Equivalent Patients With Hypercholesterolemia and Familial Hypercholesterolemia
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CKJX839A1AT01
Record Dates: First submitted 2024-07-04; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Atherosclerotic Cardiovascular Disease; Hypercholesterolemia
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Overall Cohort: Adult patients with ASCVD and hypercholesterolemia, ASCVD-RE with hypercholesterolemia, or FH, who were prescribed inclisiran in a real-world setting as per clinical practice and according to the label in Austria.

SUMMARY:
This was a descriptive, non-interventional, retrospective cohort study among patients with atherosclerotic cardiovascular disease (ASCVD) and hypercholesterolemia, ASCVD-risk equivalent (ASCVD-RE) or familial hypercholesterolemia (FH) administered inclisiran in a real-world setting in Austria.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were 18 years or older.
* Signed informed consent was obtained.
* Patients who received at least one inclisiran injection in the identification period.
* Patients with at least one diagnosis of ASCVD, ASCVD-RE or FH diagnosis prior to index date.
* Patients with at least one low-density lipoprotein cholesterol (LDL-C) measurement of 70 milligrams per deciliter (mg/dL) or greater, within 6 months prior to index date.

ASCVD was defined as previous diagnosis of coronary artery disease (CAD), peripheral artery disease (PAD) or cerebrovascular disease (CVD).

ASCVD-RE was defined as: no previous diagnosis of ASCVD at any time on the patient chart and they met at least one of the following criteria:

* Diagnosis of type II diabetes mellitus (T2DM).
* Diagnosis of type I diabetes mellitus (T1DM) of long duration (greater than 20 years).
* 10-year risk of 20% or greater by Framingham risk score.

Exclusion Criteria:

• None.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients who Received Inclisiran Dose 2 and 3 Within Specified Time Intervals | Up to 26 months
  Time intervals:
  * Time from Dose 1 to Dose 2: 5 months or less.
  * Time from Dose 2 to Dose 3:
    * Less than 6 months.
    * Between 6 months and 9 months.
    * Greater than 9 months.

SECONDARY OUTCOMES:
Percentage of Patients Taking Different Concomitant Lipid Lowering Therapy (LLT) at Index Date | Day 1 of Month 6
  Index date was defined as the date of first administration of inclisiran.
Percentage of Patients who Received Inclisiran Doses Within Specified Time Intervals | Up to 26 months
  Time intervals:
  * Time from Dose 1 to Dose 2:
    * Less than 3.5 months.
    * Between 3.5 and 5 months.
    * Greater than 5 months.
  * Time from Dose 2 to Dose 3:
    * Less than 6 months.
    * Between 6 and 7 months.
    * Between 7 and 8 months.
    * Between 8 and 9 months.
    * Greater than 9 months.
Gender | Baseline
Race | Baseline
Smoking Status | Baseline
  Patient smoker status:
  * Non-smoker
  * Current smoker
  * Past smoker
  * Unknown
Physical Activity | Baseline
  Physical activity was classified as intense, light, moderate, or unknown.
Prescribing Physician Specialty | Baseline
Age | Baseline
Weight | Baseline
Height | Baseline
Body Mass Index | Baseline
Blood Pressure | Baseline
  Blood pressure: systolic and diastolic.
Percentage of Male Patients by Age Group | Baseline
  Age groups:
  * Less than 15 years old.
  * 15 to 19 years old.
  * 20 to 29 years old.
  * 30 to 39 years old.
  * 40 to 49 years old.
  * 50 to 59 years old.
  * 60 years or older.
Percentage of Female Patients by Age Group | Baseline
  Age groups:
  * Less than 15 years old.
  * 15 to 19 years old.
  * 20 to 29 years old.
  * 30 to 39 years old.
  * 40 to 49 years old.
  * 50 to 59 years old.
  * 60 years or older.
Percentage of Patients Categorized by Comorbidities | Baseline
Cholesterol | Baseline
  Cholesterol included:
  * Low-density lipoprotein cholesterol.
  * High-density lipoprotein cholesterol.
  * Non-high-density lipoprotein cholesterol.
  * Total cholesterol.
Triglycerides | Baseline
Apolipoprotein B | Baseline
Glycated hemoglobin | Baseline
Lipoprotein(a) | Baseline
Creatinine | Baseline
Alanine Aminotransferase | Baseline
Aspartate Aminotransferase | Baseline
Alkaline phosphatase | Baseline
Percentage of Patients With Procedures | Baseline
Percentage of Atherosclerotic Cardiovascular Disease (ASCVD) Patients Categorized by Qualifying Diagnosis | Baseline
  Qualifying diagnoses were coronary artery disease (CAD), peripheral artery disease (PAD), and cerebrovascular disease (CVD).
Percentage of ASCVD-risk Equivalent Patients Categorized by Qualifying Criteria | Baseline
  Qualifying Criteria:
  * Type II diabetes mellitus.
  * Framingham risk score of 20% or greater.
  * Type I diabetes mellitus of for more than 20 years.
Percentage of Patients Categorized by Lipid Lowering Therapies (LLTs) Prior to Index Date | Up to 6 months pre-index date
  Index date was defined as the date of first administration of inclisiran.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States